CLINICAL TRIAL: NCT04876300
Title: Predicting the Cumulative Live Birth Rate Further Ovarian Stimulation by Highly Purified Human Menotropin HP-hMG. A Multicentre, Retrospective Study
Brief Title: MEDAM (Menopur Retrospective Data prograM)
Acronym: MEDAM
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000376
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-11

CONDITIONS: Infertility, Female
Keywords: Menotropin; HP-hMG
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Menotropin Cohort
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — All directions for medication usage were solely at the discretion of the investigator in accordance with their usual routine clinical practice and are assumed to be consistent with the national prescribing information of the medicinal product in the country in which the study will take place.

SUMMARY:
French, non-interventional, retrospective, multicentric analysis of patients who have undergone a controlled ovarian stimulation (COS) for in-vitro fertilization (IVF)/ intracytoplasmic sperm injection (ICSI). The main objective is to determine the cumulative live birth rate with highly purified menotropin (HP-hMG) which is defined as the occurrence of live birth per started COS, further to transfer of fresh and frozen embryos generated from the same COS.

ELIGIBILITY:
Inclusion Criteria:

- Patient undergoing a COS with HP-hMG for IVF/ICSI cycle from a French data registry between 2009 to 2016

Exclusion Criteria:

* Ovulation inductions
* Intra-uterine inseminations
* Fertility preservations
* Oocyte donations

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Adult females who underwent COS treatment with Menotropin during 2009 to 2016.
Study Population: Adult women, fitting the inclusion/exclusion criteria, who were prescribed Menotropin during 2009 to 2016 for COS in a treatment of infertility will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 11488 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Cumulative live birth rate (cLBR) | At delivery
  Defined as the occurence of live birth per started COS, further to transfer of fresh and frozen embryos generated from the same COS.

SECONDARY OUTCOMES:
Initial dose of Menotropin treatment per IVF cycle (IU) | At Day 1 of Menotropin stimulation up to Day 20 of Menotropin stimulation during 2009 to 2016
Total dose of Menotropin treatment per IVF cycle (IU) | At Day 1 of Menotropin stimulation up to Day 20 of Menotropin stimulation during 2009 to 2016
Total days of Menotropin treatment (per IVF cycle) | Up to end of the ovarian stimulation treatment (up to 20 days) during 2009 to 2016
  Duration of treatment (in days) with Menotropin of patients will be reported.
Dose adjustment of Menotropin in IU | At Day 1 of Menotropin stimulation up to Day 20 of Menotropin stimulation during 2009 to 2016
Type of gonadotropin-releasing hormone (GnRH) protocols used for Luteinizing Hormone (LH) surge suppression (with in particular long and short agonist, and antagonist) | At the day of the first GnRH administration during the ovarian stimulation treatment (up to 20 days) in 2009 to 2016
  Gonadotropin-releasing hormone protocols with in particular long and short agonist, and antagonist.
Total days of LH surge suppression protocol | From Day 1 up to the last day of GnRH analogues administration during 2009 to 2016
  Gonadotropin-releasing hormone protocols with in particular long and short agonist, and antagonist.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (9):
- France (9):
  - Ferring investigational site, Bondy
  - Ferring investigational site, Clamart
  - Ferring investigational site, Créteil
  - Ferring investigational site, Le Chesnay
  - Ferring investigational site, Lens
  - Ferring investigational site, Lyon
  - Ferring investigational site, Marseille
  - Ferring investigational site, Nice
  - Ferring investigational site, Rennes